CLINICAL TRIAL: NCT00171236
Title: Efficacy and Safety of Fluvastatin in Children With Heterozygous Familial Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CXUO320B2301
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2005-09

CONDITIONS: Heterozygous Familial Hypercholesterolemia; Mixed Dyslipidemia
Keywords: Heterozygous familial hypercholesterolemia; mixed dyslipidemia
MeSH Terms: interventions — Fluvastatin

INTERVENTIONS:
Drug: Fluvastatin

SUMMARY:
The purpose of the study is to assess the safety and efficacy of fluvastatin in children diagnosed with heterozygous familial hypercholesterolemia

ELIGIBILITY:
Inclusion Criteria:

* 10-16 years old Heterozygous familial hypercholesterolemia

Exclusion Criteria:

* Homozygous familial hypercholesterolemia Pregnant or lactating females Major surgery during the six month prior study

Other protocol defined inclusion and exclusion criteria may apply

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2001-10; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Basel, Switzerland